CLINICAL TRIAL: NCT07208708
Title: Patient Satisfaction With At-home Dental Bleaching Using Orthodontic Retainers With Different Margin Designs: a Randomized Equivalence Clinical Trial.
Brief Title: Patient Satisfaction With At-home Dental Bleaching Using Orthodontic Retainers With Different Margin Designs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Isabel Giráldez de Luis, PhD DDS, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: URJC_IDIBO_4
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Patient Satisfaction; Bleaching Efficacy; Tooth Sensitivity; Gingival Irritation
Keywords: dental bleaching; color change; hydrogen peroxide; clinical trials
MeSH Terms: conditions — Patient Satisfaction; Dentin Sensitivity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scalloped margin retainer (Active Comparator)
  Interventions: Other: Scalloped margin retainer
- Straight margin retainer (Experimental)
  Interventions: Other: Straight orthodontic retainer

INTERVENTIONS:
Other: Scalloped margin retainer — Patient satisfaction was assessed during 2 weeks of whitening with a scalloped orthodontic retainer. Colour change, TS and IG were also measured. No studies have evaluated the effect of different margin designs in orthodontic retainers used in for tooth bleaching. Therefore, the present study aimed to clinically assess the impact of scalloped and straight margin design in orthodontic retainers employed for at-home bleaching, considering patient satisfaction, bleaching efficacy, tooth sensitivity (TS), and gingival irritation (GI).
  Arms: Scalloped margin retainer
Other: Straight orthodontic retainer — Patient satisfaction was assessed during two weeks of whitening with a straight orthodontic retainer. Colour change, TS and IG were also measured. No studies have evaluated the effect of different margin designs in orthodontic retainers used in for tooth bleaching. Therefore, the present study aimed to clinically assess the impact of scalloped and straight margin design in orthodontic retainers employed for at-home bleaching, considering patient satisfaction, bleaching efficacy, tooth sensitivity (TS), and gingival irritation (GI). The null hypotheses were that no significant differences would be observed in: (1) patient satisfaction, (2) bleaching efficacy, (3) tooth sensitivity, and (4) gingival irritation, when different margin designs are used in orthodontic retainers for at-home tooth bleaching.
  Arms: Straight margin retainer

SUMMARY:
This randomized single-blind, split-mouth clinical trial evaluated patient satisfaction with at-home dental bleaching using orthodontic retainers with different margin designs, as well as bleaching efficacy, tooth sensitivity (TS), and gingival irritation (GI).

DETAILED DESCRIPTION:
The objective of the study will be to clinically evaluate patient satisfaction, as well as the effectiveness of colour change, tooth sensitivity and gingival irritation with home whitening using 10% carbamide peroxide performed with orthodontic retainers with different cut-outs. Forty patients will be selected to receive home teeth whitening with a straight or scalloped retainer on each half-arch (n=40). The whitening procedure will be performed with 10% carbamide peroxide (Pola Night 10%) for 2 hours over 14 days. Patient satisfaction will be assessed weekly for two weeks through a series of questions using the Visual Analogue Scale (VAS 0-10). Colour will be assessed initially, weekly for two weeks and 1 month after completion of whitening, using the subjective VITA Classical scale, VITA Bleachedguide 3D-MASTER and the objective VITA Easyshade spectrophotometer. The intensity and risk of tooth sensitivity and gingival irritation will be recorded on the Visual Analogue Scale (VAS 0-10). Patient satisfaction will be assessed using the paired Student's t-test. The colour change between the groups will be compared using the paired Student's t-test. The absolute risk of tooth sensitivity and gingival irritation in both groups will be compared using the McNemar test. The intensity of tooth sensitivity and gingival irritation will be analysed using the Student's t-test for paired samples. The significance level will be 5% in all statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Completed of orthodontic treatment with Invisalign aligners (Align Technology Inc., CA, USA); willingness to undergo tooth bleaching as a complementary procedure; and current use of clear retainers. Additional criteria included age of ≥18 years of age, good general and oral health, and provision of informed consent. Eligible participants also needed anterior teeth free from carious and periodontal disease, with canines of shade A2 or darker on the VITA Classical scale (VITA Zahnfabrik, Bad Säckingen, Germany) and a Whiteness Index for Dentistry (WID) value ≤15.

Exclusion Criteria:

* History of previous bleaching; self-reported tooth sensitivity; continuous use of analgesics or anti-inflammatory drugs; pregnancy or breastfeeding; and deleterious habits such as bruxism or smoking. Participants with anterior teeth presenting fixed orthodontic appliances, attachments, restorations, endodontic treatment, color changes due to tetracyclines or fluorosis, or visible enamel cracks were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | 2 weeks
  Patient satisfaction was assessed daily using a Visual Analog Scale (VAS, 0-10) consisting of nine questions was provided to Participants completed a satisfaction diary independently throughout the 2-week bleaching period, without evaluator interference or time restrictions. The scale ranged from 0 (no problem/very good) to 10 (maximum problem/very bad), with participants marking a vertical line corresponding to their perception.

SECONDARY OUTCOMES:
Bleaching efficacy | 2 weeks
  Tooth color was evaluated at baseline and after treatment using both subjective and objective methods. Subjective evaluation was performed with the VITA Classical and VITA Bleachedguide 3D-MASTER shade guides. Objective evaluation was carried out with the VITA Easyshade spectrophotometer (Vita Zahnfabrik) using the CIELab* color system.
Tooth sensitivity | 2 weeks
  Was assessed using a 10-point Visual Analog Scale (VAS), where 0 indicated no sensitivity and 10 indicated severe sensitivity
Gingival irritation | 2 weeks
  Was assessed using the same methodology as TS, with VAS ranging from 0 (no irritation) to 10 (severe irritation)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No